CLINICAL TRIAL: NCT01865942
Title: Surgical Spinal Decompression of Metastatic Spinal Cord Compression, Minimal Access Versus Open Surgery. A Randomized Clinical Trial.
Brief Title: Surgical Spinal Decompression of Metastatic Spinal Cord Compression, Minimal Access Versus Open Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Søren Schmidt Morgen, Medical doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2011-050
Record Dates: First submitted 2013-04-04; First posted 2013-05-31 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Spinal Metastases
Keywords: spinal metastases; spine surgery; metastatic spinal cord compression; EQ-5D; HRQOL
MeSH Terms: conditions — Spinal Cord Compression | interventions — Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open surgery (Active Comparator): One arm receives open surgery. In our department open surgery is considered as the standard procedure since all spine surgeons are preforming this operation.
  Interventions: Procedure: open surgery
- Minimal access surgery (Active Comparator): We compare to well-known types of surgery for metastatic spinal cord compression. The other arm receive open surgery. In our department minimal access surgery is considered as a standard procedure but it is not preformed by all spine surgeons.
  Interventions: Procedure: Minimal access surgery

INTERVENTIONS:
Procedure: open surgery — The to surgical procedures are individually well know, but the outcome of the procedures in respect to perioperative bleeding and change in quality of life has to our knowledge not been compared.
  Arms: open surgery
Procedure: Minimal access surgery — The to surgical procedures are individually well know, but the outcome of the procedures in respect to perioperative bleeding and change in quality of life has to our knowledge not been compared.
  Arms: Minimal access surgery

SUMMARY:
The investigators wish to evaluate the effect of minimal access spinal surgery compared to traditional open surgery spinal surgery in patients with metastatic spinal cord compression.

Minimal access surgery has been shown to bee less damaging for the tissue compared to traditional open surgery and also cause fewer wound complications, the investigators expect the above could have impact in a vulnerable patient group like patients with metastatic spinal cord compression.

DETAILED DESCRIPTION:
Surgical Spinal Decompression of Metastatic Spinal Cord Compression, Minimal Access Versus Open Surgery. A Randomized Clinical Trial

Purpose To investigate the effect of minimal access spine surgery (MASS) compared with conventional open surgery in the treatment of patients with metastatic spinalcord compression (MSCC).

Hypotheses The group of patient's receiving MASS will have better improvement in quality after surgery compared to the group that will receive traditional open surgery. The MASS patient group will have reduction in per-operative bleeding and less wound complications needing surgical revision compered to the group of patients receiving open or traditional surgery.

Primary outcome Perioperative bleeding.

Secondary outcomes Quality of life and incidence of revision surgery.

Material and method A randomised controlled trial with a 1-year follow up will be conducted.

Sample size From previous studies and based patient files it is calculated that the mean blood loss during open surgery is 1500 ml (standard deviation 750 ml). A clinical relevant reduction in blood loss will be 400 ml corresponding to one unit of packed red blood cells.

With a significance level of 5% and a power of 80% a total of 62 patients have to be included in the study.

Most studies using QLQ-C30 as a measurement for health related quality of life (HRQL) in randomized comparison of treatment modalities in cancer patients have included between 100 and 200 patients. This includes studies where both QLQ-C30 and EQ-5D have been used. EQ-5D is widely used as a generic measurement of HRQL.

62 patients will be randomly allocated to receive either minimal invasive or open surgery. Inclusion criteria are patients with spinal metastases at level Th5-L3 who are candidates for surgery. Exclusion criteria are: Tokuhashi score ≤ 4, preoperative presumptions that something else than pedicle screws would be needed, potentially the need for sacral or iliosacral instrumentation, and patients who need more radical treatment. The QLQ-C30 (Quality of Life Cancer) will be assessed since this instrument is especially developed for use in cancer patients and will be used as a clinical measure.

Outcome measure on bleeding will be recorded during the operation. Outcome measures on quality of life will be estimated with QLQ-C30, EQ-5D and VAS-pain score. This will be recorded before operation, by time of discharge, 6 weeks and 3, 6 and 12 months after the operation. Records on wound complications leading to an intervention of revision-surgery, antibiotics or other procedures are registered at the same follow up times.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic spinal cord compression with a metastasis from Th5-L3 Tokuhashi above 4

Exclusion Criteria:

* Need for radical treatment and not only palliative
* Need for surgical stabilization in a region lower then L3

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Bleeding | intraoperative
  The investigators compare the bleeding for each treatment modality during the operation.

SECONDARY OUTCOMES:
Health related quality of life measured with questionnaire EQ-5D and QLQ-C30 | before intervention and six months follow up
  The EORTC EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status.
  The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Schmidt Morgen, MD, Principal Investigator — Spine Section, Department of Orthopedic Surgery, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Rodriguez-Vela J, Lobo-Escolar A, Joven-Aliaga E, Herrera A, Vicente J, Sunen E, Loste A, Tabuenca A. Perioperative and short-term advantages of mini-open approach for lumbar spinal fusion. Eur Spine J. 2009 Aug;18(8):1194-201. doi: 10.1007/s00586-009-1010-0. Epub 2009 Apr 28. PMID 19399538
- [Background] Falicov A, Fisher CG, Sparkes J, Boyd MC, Wing PC, Dvorak MF. Impact of surgical intervention on quality of life in patients with spinal metastases. Spine (Phila Pa 1976). 2006 Nov 15;31(24):2849-56. doi: 10.1097/01.brs.0000245838.37817.40. PMID 17108840
- [Background] Kim KT, Lee SH, Suk KS, Bae SC. The quantitative analysis of tissue injury markers after mini-open lumbar fusion. Spine (Phila Pa 1976). 2006 Mar 15;31(6):712-6. doi: 10.1097/01.brs.0000202533.05906.ea. PMID 16540878
- [Background] Ringel F, Stoffel M, Stuer C, Meyer B. Minimally invasive transmuscular pedicle screw fixation of the thoracic and lumbar spine. Neurosurgery. 2006 Oct;59(4 Suppl 2):ONS361-6; discussion ONS366-7. doi: 10.1227/01.NEU.0000223505.07815.74. PMID 17041505